CLINICAL TRIAL: NCT03563768
Title: Evaluation of the Strategy of "One-stop" Endovascular Treatment for Concomitant Coronary Artery Disease and Aortic Atherosclerotic Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Yi-Da Tang, Clinical professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-2-4032
Record Dates: First submitted 2018-06-10; First posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Coronary Artery Disease; Aortic Atherosclerotic Disease
Keywords: coronary artery disease; aortic atherosclerotic disease; one-stop; endovascular aortic repair; percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One-stop strategy group (Experimental): Percutaneous coronary intervention (PCI) will be performed on the same operating table immediately after the endovascular aortic repair (EVAR)
  Interventions: Procedure: One-stop strategy group
- Staging strategy group (No Intervention): PCI will be performed several days after EVAR

INTERVENTIONS:
Procedure: One-stop strategy group — Percutaneous coronary intervention (PCI) will be performed on the same operating table immediately after the endovascular aortic repair (EVAR)
  Arms: One-stop strategy group

SUMMARY:
The study is a prospective, randomized, controlled, exploratory trail to evaluate the strategy of "one-stop" endovascular treatment for concomitant coronary artery disease and aortic atherosclerotic disease.

DETAILED DESCRIPTION:
60 patients will be allocated randomly in a 1:1 ratio into one-stop strategy group or staging strategy group. In one-stop strategy group, percutaneous coronary intervention (PCI) will be performed on the same operating room immediately after the endovascular aortic repair (EVAR); In staging strategy group, PCI will be performed several days after EVAR. The safety and effectiveness will be assessed between two groups 1 year after the operation. The economic index will be evaluated as well as.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 years to 75years, male or female;
* Aortic atherosclerotic disease with indication of EVAR;
* Coronary heart disease with indication of PCI;
* Provided informed consent.

Exclusion Criteria:

* Acute aortic dissection
* Acute coronary syndrome
* Dysfunction of coagulation system
* Patients with gastrointestinal hemorrhage
* Known allergy to contrasts or antiplatelet drugs
* Renal dysfunction (GFR≤60ml/min)
* Patient with multi-branch coronary preferred CABG

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-06-30 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Perioperative major bleeding (BARC≥3 grade) | 12 months

SECONDARY OUTCOMES:
Difference of operative success rate between two groups | 12 months
Difference of incidence of all-cause death between two groups | 12 months
Difference of incidence of myocardial infarction between two groups | 12 months
Difference of incidence of rupture of aorta between two groups | 12 months
Difference of incidence of bleeding events (BARC 2 grade) between two groups | 12 months
Difference of incidence of pseudoaneurysm between two groups | 12 months
Difference of incidence of Stent thrombosis between two groups | 12 months
Composite of average in-patient time and average cost during hospitalization | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Da Tang, MD, PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Chinese Academy of Medical Sciences, Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No